CLINICAL TRIAL: NCT04890574
Title: An Open Label Pilot Study to Evaluate the CellMist™ System in the Treatment of Deep Second Degree (IIoB) Burn Injuries With Autologous Skin Cells
Brief Title: CellMist™ Autologous Cells to Treat Deep Second-Degree Burns
Acronym: CELLMIST1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RenovaCare, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC12302017
Record Dates: First submitted 2021-04-29; First posted 2021-05-18 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Burns; Burns Second Degree; Burns Deep Second Degree
Keywords: Cell Therapy; Burn Injury
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: This is a prospective, single arm, open label non-randomized safety and device feasibility study.
Masking Description: This is a prospective, single arm, open label non-randomized safety and device feasibility study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: CellMist™ System — Open Label, Safety and Feasibility

SUMMARY:
The overall purpose of this study is to evaluate the safety of the CellMist™ System in the treatment of deep second degree burns (II°B) in a prospective, multicenter, feasibility pilot study.

DETAILED DESCRIPTION:
Patients between the ages of 18 and 65 years of age inclusive with a ≤ 30% Total Body Surface Area (TBSA) that requires surgical or enzymatic debridement and split thickness skin grafting (STSG) on any body surface excluding the face, joints, perineum and hands will be considered for participation in this study. CellMist™ solution (autologous epidermal and dermal cells) will be administered, via the System Skin Gun™, will be evenly distributed to aid in burn healing. Healing, pain and treatment-related adverse events will be evaluated at follow-up visits. Data concerning safety of the CellMist™ System will be collected. Safety will be evaluated in terms of treatment and serious related adverse events.

Each subject will participate in up to 9 total visits (screening, treatment and 7 follow-up study visits) over a period of 52 weeks. Up to 14 subjects will be enrolled and treated within this at up to 4 institutions.

ELIGIBILITY:
Inclusion Criteria:

1. Is between 18 and 65 years of age inclusive;
2. Has at least one discrete deep second degree (II°B) thermal burn injury (≤ 30% Total Body Surface Area (TBSA)) that requires surgical or enzymatic debridement and split thickness skin grafting (STSF) on any body surface excluding the face, joints, perineum and hands;
3. Agrees to abstain from any other surgical treatment of the wound(s) for the duration of the study unless determined by the Principal Investigator to be medically necessary;
4. Treatment with CellMist™ occurs with 7 days of burn injury;
5. Demonstrates (as determined by the Principal Investigator) the ability and willingness to follow the requirements of the protocol;
6. Understand the full nature and purpose of the study and provides voluntary written informed consent -

Exclusion Criteria:

1. Is pregnant or does not agree to use acceptable contraception methods for the duration of their participation in the clinical trial (latter applies to women and men of child bearing potential);
2. Is breast feeding;
3. Has a pre-existing local and/or systemic bacterial infection that requires antibiotic treatment for more than 2 days prior to study treatment;
4. Demonstrates an anesthesia risk that (as determined by the Principal Investigator) prohibits treatment
5. Body Mass Index (BMI) ≥ 39;
6. The burn(s) at the target treatment area(s) results from chemical, electrical or radiation exposure;
7. Has full thickness (III°) burns TBSA ≥ 20%
8. Has comorbidities and/or medications and/or health status that (as determined by the Principal Investigator) could result in poor cell isolation and/or poor wound healing (e.g., uncontrolled and/or significant diabetes (≥8% HbA1c by medical record), peripheral vascular disease, active malignancy or treatment (other than surgery) of malignancy within the past 3 months, autoimmune disease, renal failure (glomerular filtration rate <60mL/minute) and/or systemic steroid usage);
9. Known hypersensitivities to trypsin, collagenase, or GentLyase (dispase);
10. Has a medical condition that would make life expectancy < 12 months;
11. Is currently participating in another prospective investigational clinical trial;
12. Does not agree to abstain from enrolling in any other study for the duration of this study;
13. Gram staining of SkinGun™ cell suspension output shows excessive microbial bioburden (≥ 200 microbial particles/field)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
All Adverse Events | We will be evaluating all adverse events reported for the period from enrollment through the final visit which will be 12 months
  All Adverse Events will be reported, recorded and analyzed which occur from the time Informed Consent is given through the conclusion of the study. We will be looking at ; Incidence, Severity, Expectedness, Duration, Treatment, and the Relationship to Device for each Adverse Event reported.
Secondary Surgical Interventions | The evaluation will include all reported secondary surgical interventions for the period from enrollment and up to 12 months
  We will be evaluating and analyzing all secondary surgical interventions required to treat the intended target wound. A secondary surgical intervention may include debridement, biopsy, identification of an infectious pathogen, split thickness skin graft, etc...

CONTACTS AND LOCATIONS:
Locations (1):
- Washington MedStar Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided